CLINICAL TRIAL: NCT02594306
Title: Brain Electrophysiological Study(EEG/ERP) on Opiate Addicts Treating by Bilateral NAc/ALIC Deep Brain Stimulation
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Tang-Du Hospital (Other)
Responsible Party: Principal Investigator, Guodong Gao, Neurosurgery Department, Tang-Du Hospital
Allocation: Non-Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: EEG/ERP and drug addiction
Record Dates: First submitted 2015-10-14; First posted 2015-11-03 (Estimated); Last update posted 2016-02-19 (Estimated); Status verified 2016-02

CONDITIONS: Substance-Related Disorders
Keywords: drug addiction; Heroin; craving; event related potential; crystal methamphetamine
MeSH Terms: conditions — Substance-Related Disorders | interventions — Deep Brain Stimulation; Microelectrodes

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- Non operation (Experimental): Recording the event related potential of drug addicts when they receive the stimulus of Emotional pictures stimulation system.
  Interventions: Device: Emotional pictures stimulation system
- Deep brain stimulation (Experimental): Recording the event related potential after the deep brain stimulation operation.Recording the local field potential of drug addiction people when we conduct a test of adjacent contact stimulation in the deep brain stimulation operation. Recording the waveform of bilateral NAc/ALIC after puting the microelectrodes into bilateral nucleus accumbens and anterior limb of the internal capsule
  Interventions: Device: Emotional pictures stimulation system; Procedure: Deep brain stimulation; Procedure: adjacent contact stimulation; Procedure: microelectrode
- Standard Control (Active Comparator): Recording the event related potential of normal people when they receive the stimulus of emotional pictures stimulation system.
  Interventions: Device: Emotional pictures stimulation system

INTERVENTIONS:
Device: Emotional pictures stimulation system — Emotional pictures stimulation system is component of neutral and drug-related images.
Procedure: Deep brain stimulation — Deep brain stimulation of bilateral NAc/ALIC
  Arms: Deep brain stimulation
Procedure: adjacent contact stimulation — The electrode of deep brain stimulation has four contacts.We stimulate one contact,and record the local field potential of other contacts.
  Arms: Deep brain stimulation
Procedure: microelectrode — We put the microelectrodes into bilateral nucleus accumbens and anterior limb of the internal capsule,to record the waveform of bilateral NAc/ALIC.
  Arms: Deep brain stimulation

SUMMARY:
Drug addiction is compulsive and spontaneous drug-taking behavior which is characterized by non-medical usage, long and repeated exposure to addictive drugs and gradually increasing drug-taking dosage and frequency,and become a main threat against human being's public health, economic development and social safety.

DETAILED DESCRIPTION:
Effective treatments for severe drug addiction are limited. China centers employing compulsory detoxification, reported a 3 year abstinence rate of only 15%. For the methadone maintenance therapy, relapse often occurs promptly after cessation of methadone. A Malaysian reports about taking naltrexone or buprenorphine treating,showed average relapsed time of 2 or 3 months,respectively.

Assessment for psychological craving degree of addiction patients is also a difficult thing.

ELIGIBILITY:
Inclusion Criteria:

1. Age between 18 and 65 years of age, male or female；
2. Opiate addictive over 3 years；
3. Physical detoxification completed（keep abstinent for at least 7 days，acute abstinent syndrome disappeared，morphine urinalysis and naloxone test showed negative)；
4. No obvious neuropsychiatry and personality disorders；
5. No severe infectious disease；
6. Good compliance and be able to complete follow up；
7. General health is good，no severe liver、kidney、heart and lung disease；
8. Informed consent issued

Exclusion Criteria:

1. Severe cognitive disorders（MMSE scale: illiteracy≤17，primary school≤20，secondary school or above≤24）,bad compliance because of dementia,unable to issue the informed content；
2. History of severe neuropsychiatric disease；
3. Epilepsy；
4. severe liver、kidney、heart and lung disease, severe hypertension and severe orthostatic hypotension；
5. Malignant tumor；History of brain trauma；Pregnant female；
6. Patients are taking part in other clinical trials in recent 3 months；
7. Being deem as unfit for the trials by researcher.

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 20 (Estimated)
Dates: Start 2015-10; Primary Completion 2016-11 (Estimated); Study Completion 2016-11 (Estimated)

PRIMARY OUTCOMES:
Event related potentials(ERPs) | Day 3
  Event related potentials include late positive potential（LPP),P300,mismatch negativity(MMN) and N400.Recording the event related potential when people receive the stimulus of emotional pictures stimulation system.

SECONDARY OUTCOMES:
local field potential(LFP) | in surgery,3 days after surgery
  Recording the LFP of DBS group without any stimulation and stimulate one contact in surgery and 3 days after surgery.
the 13-item obsessive compulsive drug use scale(OCDUS) | day 3
Opiate Addiction Severity Inventory(OASI) | day 3
participants' craving for opioid drugs (VAS) | day 3
  The 10-point visual analog scale(VAS)will be utilized at day 3.
The Symptom Checklist-90(SCL-90) | day 3
  The Symptom Checklist-90(SCL-90) is used to evaluate general status.
Self-Rating Depression Scale(SDS) | day 3
  Self-Rating Depression Scale(SDS) is used to evaluate depression symptom.
Yale-Brown Obsessive Compulsive Scale(Y-BOCS) | day 3
  Yale-Brown Obsessive Compulsive Scale(Y-BOCS) is used to evaluate obsessive compulsive symptom.
The Eysenck Personality Questionnaire(EPQ) | day 3
The Wechsler Memory Scale(WMS) | day 3

CONTACTS AND LOCATIONS:
Overall Officials: Guo-dong Gao, M.D., Study Chair — Department of neurosurgery, Tangdu Hospital
Locations (1):
- Department of neurosurgery, Tangdu Hospital, Xi'an, Shaanxi, China